CLINICAL TRIAL: NCT00917826
Title: A Phase II Trial of Low-Dose Arginine Butyrate and Ganciclovir/Valganciclovir in EBV(+)Lymphoid Malignancies
Brief Title: Study of Arginine Butyrate and Ganciclovir/Valganciclovir in EBV(+) Lymphoid Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: HemaQuest Pharmaceuticals Inc. (Industry)
Collaborators: Boston University (Other)
Responsible Party: Susan Perrine, M.D. Chief Scientific Officer, VP Clinical Affairs, HemaQuest Pharmaceuticals Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2 L-D AB
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: EBV Lymphomas; Lympho-proliferative Diseases
MeSH Terms: interventions — arginine butyrate; Ganciclovir; Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arginine Butyrate + Ganciclovir/Valganciclovir (Experimental)
  Interventions: Drug: Arginine Butyrate; Drug: Ganciclovir; Drug: Valganciclovir

INTERVENTIONS:
Drug: Arginine Butyrate — 1,000 mg/kg/day administered IV over 24 hours/day for 5 days (Days 1-5 of each 21 day cycle)
  Other Names: HQK-1004
Drug: Ganciclovir — 5 mg/kg administered IV over 1 hour (Days 1-5 of each 21 day cycle)
Drug: Valganciclovir — 900 mg BID for 16 days (Days 6-21 of each 21 day cycle)

SUMMARY:
The purpose of this study is to assess whether administration of Arginine Butyrate + ganciclovir/valganciclovir for up to three 21-day cycles is tolerable, and results in partial or complete responses in patients with EBV(+) lymphoid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 3 years. (No dosing or adverse event data are currently available on the use of valganciclovir in patients < 16 years of age.)
* Life expectancy of > 3 months.
* ECOG Performance Status 0-2 or Karnofsky Performance Scale ≥ 60%.
* Baseline (untransfused) HbF level > 2%
* Normal organ and marrow function defined as: (i) absolute neutrophil count of ≥ 1,000/µL. (ii) platelets ≥ 50,000/ µL. (iii) total bilirubin of ≤ 2.0 x upper limit of normal. (iv) AST (SGOT)/ALT(SGPT) of ≤ 2.0 x institutional upper limit of normal. (v) creatinine within normal range for institution.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Able and willing to give informed consent.

Exclusion Criteria:

* Patients that have received chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entry, or those who have not recovered form adverse events due to agents administered 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Arginine Butyrate, ganciclovir or valganciclovir.
* Patients who have an acute myocardial infarction or onset of atrial fibrillation within the past 6 months.
* Uncontrolled intercurrent illness including, but not limited to , ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Tumor impinging on an organ or anatomical structure deemed critical by the investigator.
* Pregnant women.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Response Rate (using Revised Response Criteria for Malignant Lymphoma, Cheson et al., JCO 2007) | Every three weeks. If a response is recorded evaluation continues until an objective determination of disease progression is made (assessment may continue after treatment is discontinued.)

SECONDARY OUTCOMES:
Progression Rate (using Revised Response Criteria for Malignant Lymphoma, Cheson et al., JCO 2007) | Every three weeks. If a response is recorded evaluation continues until an objective determination of disease progression is made (assessment may continue after treatment is discontinued.)
Safety as assessed by (1) adverse events, (2) laboratory values (3) vital signs (4) physical exam | Up to three 21-day cycles. If a response is recorded evaluation continues until an objective determination of disease progression is made (assessments may continue after treatment is discontinued.)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Lerner, M.D., Principal Investigator — Boston University School of Mediciine
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States